CLINICAL TRIAL: NCT04953416
Title: Evaluation of Safety and Performance of Fractional Non-ablative Laser for the Treatment of Hair Loss - A Pilot Study
Brief Title: Fractional Non-ablative Laser for the Treatment of Hair Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-M22-ResurFX-19-01
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Scalp treatment with ResurFX (Experimental)
  Interventions: Device: 1565nm non ablative fractional laser

INTERVENTIONS:
Device: 1565nm non ablative fractional laser — The ResurFX module contains Erbium:Glass Fiber Laser Technology with wavelength of 1565 nm, which is transferred to the ResurFX handpiece via a fiber.
  Other Names: ResurFX by Lumenis Ltd.

SUMMARY:
This is a single center, prospective, open label clinical trial with before-after study design. The study is designed to evaluate the feasibility of hair growth in female and male pattern hair loss (androgenic alopecia, telogen effluvium, and alopecia areata) using a fractional non-ablative 1565nm ResurFX module.

DETAILED DESCRIPTION:
This is a single center, prospective, open label clinical trial with before-after study design. The study is designed to evaluate the feasibility of hair growth in female and male pattern hair loss (androgenic alopecia, alopecia areata) using a fractional non-ablative 1565nm ResurFX module.

This study will include up to 13 visits at the clinic: screening; at least 5 and up to 10 treatment (Tx) visits 14+/-3 days apart, and follow up (FU) visits at 1 and 3 months (each can be +/-7 days out of window) after the last treatment session. See Figure 3: Study Design for an illustration of the study design, for a summary of the study procedures and Table 1 for the schedule of times and events.

The study population will include up to 35 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with noticeable alopecia of the following types: androgenic alopecia, telogen effluvium and alopecia areata
* Experiencing active hair loss within the last 1 months but no longer than 5 years
* Male/Female hair pattern loss base on:

  1. Male presenting Norwood Hamilton Scale - Stage 1 and up to 4
  2. Female presenting Sinclair Grade I-IV
* Subjects in general good health
* Male and female, age 18-45 years old
* Women of child-bearing potential that agree to abstain from pregnancy or breastfeeding during the course of the study
* Women of child-bearing potential are required to use a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, NuvaRing, partner with vasectomy, Implanon or other approved devices, or abstinence) at least 3 months prior to enrollment and throughout the course of the study
* Willing to remain on the same diet/habits (per physician recommendation)
* Subject is willing and able to comply with protocol requirements and all study visits
* Subject is willing and able to provide a written informed consent

Exclusion Criteria:

* Male/Female hair pattern loss base on:

  1. Male presenting Norwood Hamilton Scale - Stage 5 and up to 7
  2. Female presenting Sinclair Grade V
* Subjects who suffer from scarring alopecia or alopecia totalis
* Women who are pregnant, lactating, or less than 6 months post-lactation completion, possibly pregnant or planning a pregnancy during the study period
* Currently participating in or recently participated in another clinical trial (within the last 90 days)
* Has photosensitivity to laser treatment

Previous/Current Alopecia Treatment

* Has used during the six months prior to screening or is currently on any of the following medications: finasteride (or any other 5α-reductase inhibitor medications), medications with anti-androgenic properties, topical estrogen, progesterone, tamoxifen, anabolic steroids, medications which can potential cause hypertrichosis, oral glucocorticoids, lithium, phenothiazines, or other medication at the discretion of the investigator
* Has used during 6 months prior to screening or is currently on Minoxidil
* Has used oral phytotherapy within 2 months prior to study

Treatment area related

* Subject who color (any type of dye) their hair less than 2 weeks prior to treatment and can't withhold dying their hair during the course of the treatment period.
* Has any active skin infection in the scalp or scarring
* Has had hair transplants, scalp reduction, current hair weave or tattooing in the target area, which makes it difficult to perform treatment and assessments
* Has a chronic dermatological condition (eczema, psoriasis, infection, etc.) of the scalp
* Has ever received radiation therapy to the scalp

Medical Conditions

* History of cancer with the exception of (1) successfully treated basal cell or squamous cell carcinoma of the skin or (2) subjects with a history of successfully treated cancer that have been disease-free for five years (not in the treatment area)
* Any current cancer, or has had chemotherapy in the past year
* Bleeding disorders and/or using anti-platelet and anticoagulant medication
* Uncontrolled systemic disease (diabetes) or infection
* History of hypogonadism
* Has significant systemic illness
* Has a known underlying medical problem that could influence hair growth such as HIV infection, connective tissue disease, a thyroid condition, inflammatory bowel disease or other medical conditions, at the discretion of the investigator.
* Has used Accutane in the past 6 months
* Has a history of poor wound healing
* Has a history of keloid formation
* Has a history or evidence of heavy smoking (more than 1 package/20 cigarettes a day), any drug and/or alcohol abuse (over 500ml of 40% hard liquor a week) within the 12 months prior to study
* Significant concurrent illness that, in the investigator's opinion would interfere with the subject's participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Hair Density Improvement | week 0 and week 24 week follow up
  evaluate the change in hair density in the target area hair count between baseline and follow up (at 1 month following last treatment), as assessed by scalp macro-imaging.

SECONDARY OUTCOMES:
Subjective Improvement | 24 week and 32 week follow up
  Subjective global assessment of hair regrowth by subjects and the investigator at 1 and 3 months following last treatment using a 5-point improvement scale
Hair Density Improvement | week 0 and week 32 week follow up
  Change in hair density in the target area between baseline and 3 month following last treatment, as assessed by scalp macro-imaging.
Adverse events | week: 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 32
  Skin safety throughout the study as determined by the investigator by examining the post-treatment occurrences of complications and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Olga Yarish, MD, Principal Investigator — AMG clinic
Locations (1):
- AMG, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: No
As this is a feasibility evaluation we do not want to publish yet.